CLINICAL TRIAL: NCT00755079
Title: A Randomized, Double-blind, Placebo-controlled Parallel Group Trial to Determine the Effect of an Oral Beta-2 Agonist on Respiratory Muscle Strength in Spinal Cord Injury
Brief Title: Use of an Oral Beta-2 Agonist in Persons With Spinal Cord Injury
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B4162-C
Record Dates: First submitted 2008-09-15; First posted 2008-09-18 (Estimated); Results first posted 2014-07-16 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-02

CONDITIONS: Spinal Cord Injury
Keywords: spinal cord injury; beta-2 agonist; respiratory muscle strength; pulmonary function test
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Placebo Comparator): group of persons with spinal cord injury will receive blinded placebo capsule
  Interventions: Drug: placebo
- Arm 2 (Experimental): group of persons with spinal cord injury will receive blinded beta-2 adrenergic agonist capsule
  Interventions: Drug: extended release beta-2 adrenergic agonist

INTERVENTIONS:
Drug: extended release beta-2 adrenergic agonist — Albuterol extended release belongs to a class of drugs known as bronchodilators. It works in the airways by opening breathing passages and relaxing muscles.
  Arms: Arm 2
Drug: placebo — An ambiguous sheathing capsule will be placed over a lactose placebo pill. The placebo will have no effect on pulmonary function.
  Arms: Arm 1

SUMMARY:
The primary purpose of this study is to determine the effect of administration of the oral beta-2 adrenergic agonist, albuterol, on respiratory muscle strength in individuals with cervical (neck) and high thoracic (upper back) spinal cord injury and to compare findings with those obtained in a demographically matched group that will receive placebo. Participation in this study will involve 12 weeks of pharmacological intervention during which participants will be randomized to receive either oral albuterol 4mg twice daily or placebo. All investigators and study participants will be blinded to randomization by our research pharmacy. Participation in the study will require study subjects to come to our lab for the total of 2 visits (at baseline and after week 12), during which a series of tests will be performed to assess their respiratory muscle strength and pulmonary function.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Spinal Cord Injury (>1 year post-injury)
* All American Spinal Injury Association (ASIA) classifications
* High Paraplegia (level of injury T1-T6)
* Tetraplegia (level of injury C2-C8, non-ventilator dependent)

Exclusion Criteria:

* history of asthma
* uncontrolled hypertension or cardiovascular disease
* those using beta-2 adrenergic agonists
* epilepsy or seizure disorder
* hyperthyroidism
* chronic corticosteroid use
* those taking monoamine oxidase inhibitors or Tricyclic antidepressants for depression
* hypersensitivity to albuterol or any of its' delete components
* pregnancy
* use of ergogenic aids or supplements with anabolic characteristics including, but not limited to:

  * creatine monohydrate
  * anabolic steroids (e.g., testosterone)
  * growth hormone and their analogs and/or derivatives

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2007-04; Primary Completion 2012-08 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Greg Schilero, MD, Principal Investigator — VA Medical Center, Bronx
Locations (1):
- VA Medical Center, Bronx, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Control: group of persons with spinal cord injury will receive blinded placebo capsule
  placebo: An ambiguous sheathing capsule will be placed over a lactose placebo pill. The placebo will have no effect on pulmonary function.
- Active Drug: group of persons with spinal cord injury will receive blinded beta-2 adrenergic agonist capsule
  extended release beta-2 adrenergic agonist: Albuterol extended release belongs to a class of drugs known as bronchodilators. It works in the airways by opening breathing passages and relaxing muscles.
Period: Overall Study
Arm/Group | Placebo Control | Active Drug
Started | 18 | 22
Completed | 17 | 16
Not Completed | 1 | 6
Not completed — Lost to Follow-up | 1 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Placebo: group of persons with spinal cord injury will receive blinded placebo capsule
  placebo: An ambiguous sheathing capsule will be placed over a lactose placebo pill. The placebo will have no effect on pulmonary function.
- Total: Total of all reporting groups
Arm/Group | Placebo | Active Drug | Total
Number analyzed (Participants) | 17 | 16 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.24 (9.53) | 42.75 (14.74) | 42.48 (12.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 16 | 15 | 31
Region of Enrollment [Number; unit: participants]
  United States | 17 | 16 | 33

OUTCOME MEASURES:

1. Primary Outcome: Inspiratory Respiratory Muscle Strength
Description: Respiratory muscle strength as measured by maximal inspiratory and pressures at the mouth.
Time Frame: Outcome will be measured at baseline, prior to intervention, and after 12 weeks of twice daily drug treatment.
Measure: Mean (Standard Deviation); unit: cmH2O
Arm/Group | Placebo Control | Active Drug
Number analyzed (Participants) | 17 | 16
cmH2O
  Maximal Inspiratory Pressure Baseline | 82.35 (18.07) | 79.19 (29.72)
  Maximal Inspiratory Pressure 12wk Post | 85.31 (24.51) | 91.69 (32.04)

2. Secondary Outcome: Expiratory Respiratory Muscle Strength
Description: Respiratory Muscle Strength defines as Maximal expiratory muscle strength at the mouth.
Time Frame: Outcome will be measured at baseline, prior to intervention, and after 12 weeks of twice daily drug treatment.
Measure: Mean (Standard Deviation); unit: cmH2O
Arm/Group | Placebo Control | Active Drug
Number analyzed (Participants) | 17 | 16
cmH2O
  Maximal Expiratory Pressure Baseline | 84.65 (36.82) | 70.38 (35.95)
  Maximal Expiratory Pressure 12 week | 88.31 (30.12) | 77.44 (37.89)

ADVERSE EVENTS:
Arm/Group | Placebo | Active Drug
Serious Adverse Events (participants affected / at risk) | 0/18 | 1/22
Other Adverse Events (participants affected / at risk) | 0/18 | 0/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=18) | Active Drug (N=22)
Muscle Cramping (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes